CLINICAL TRIAL: NCT06026332
Title: ADSTILADRIN Early Utilization and Outcomes in the Real World Setting
Acronym: ABLE-41
Status: Recruiting | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000431
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; NMIBC; CIS; Ta/T1; BCG Unresponsive; Vesical instillation treatment
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ADSTILADRIN
  Interventions: Drug: ADSTILADRIN

INTERVENTIONS:
Drug: ADSTILADRIN — Non-interventional
  Other Names: Nadofaragene Firadenovec

SUMMARY:
Multi-center, prospective non-interventional study to collect data on the early use of Adstiladrin in the US and Israel. Data will be collected from patients and prescribing physicians in a real-world setting

ELIGIBILITY:
Inclusion Criteria:

* Prescribed and scheduled treatment with ADSTILADRIN per physician discretion or received the first instillation of ADSTILADRIN per physician discretion after 5 September 2023 but prior to site activation
* Signed and dated ICF.
* Age 18 years or older at day ICF is signed.

Exclusion Criteria:

* Currently enrolled in a clinical trial.
* Participants who have previously been treated with ADSTILADRIN in the context of a clinical trial
* Participant is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been prescribed Ferring ADSTILADRIN at the participating sites will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Whether or not a patient with CIS (with or without concomitant high-grade Ta or T1 papillary disease) achieves Complete Response (CR) at first evaluation from first ADSTILADRIN instillation | 3 months
Whether or not a patient with CIS (with or without concomitant high-grade Ta or T1 papillary disease) achieves CR at any time within 1 year from first ADSTILADRIN instillation | 1 year

SECONDARY OUTCOMES:
Duration of CR in patients with CIS (with or without concomitant high-grade Ta or T1 papillary disease) who achieve CR | Up to 2 years
High-grade recurrence-free survival | Up to 2 years
Incidence of being HGRF after one ADSTILADRIN instillation and incidence of being HGRF at 1 year from first ADSTILADRIN instillation | 1 year
Incidence of and time to cystectomy | Up to 2 years
Progression-free survival (PFS) | Up to 2 years
Overall Survival (OS) | Up to 2 years
Mortality due to bladder cancer | Up to 2 years
Prior treatments and outcomes before starting ADSTILADRIN treatment | Before starting ADSTILADRIN treatment
Number of ADSTILADRIN instillations received and time intervals between instillations | Up to 2 years
Reasons for discontinuation of ADSTILADRIN treatment | End of trial (up to 2 years)
Concomitant therapies for bladder cancer and major comorbidities | Up to 2 years
Re-treatment of non-responders with ADSTILADRIN at 3 months or when deemed appropriate by the treating physician | 3 months
Patients' caregiver experience as measured by WPAI:CG (administered at the same timepoints as the patients) | Up to 2 years
  WPAI:CG is Work Productivity and Activity Impairment, as adapted for caregiving.
Subsequent line of therapy following ADSTILADRIN discontinuation | Up to 2 years
Customized patient baseline and follow-up experience surveys (before first ADSTILADRIN instillation and before each instillation thereafter) | Before first ADSTILADRIN instillation and before each instillation thereafter
Quality of life surveys (EQ-5D-5L before first ADSTILADRIN instillation) | Before first ADSTILADRIN instillation
Customized physician surveys (at 1 month following first patient first instillation of ADSTILADRIN, or as soon as possible upon site activation, and at 12 and 24 months post first patient first instillation at each respective site) | Up to 2 years
  Domains captured will include product considerations and treatment satisfaction
Type, incidence, relatedness to ADSTILADRIN, severity grading (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0), and seriousness of adverse events collected | End of trial (up to 2 years)
Proportion of patients with pre-specified biomarker tested in the routine care setting, along with timing, type of sampling and laboratory results | End of trial (up to 2 years)
  Routine care setting e.g., Cxbladder Detec, UroVysion FISH, nuclear matrix protein 22 (NMP22) and bladder tumor antigen (BTA) tests]

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (30):
- United States (30):
  - Banner Health MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arkansas Urology, North Little Rock, Little Rock, Arkansas
  - Urology Associates of Central California, Fresno, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UF Health Surgical Specialists - Gainesville, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Urology Partners, Riverview, Florida
  - Florida Urology Partners, St. Petersburg, Florida
  - Florida Urology Partners, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Urology, Atlanta, Georgia
  - UROLOGY OF INDIANA - GREENWOOD FQ: Urology of Indiana US Uro Partners, Greenwood, Indiana
  - First Urology Research (Jeffersonville), Jeffersonville, Indiana
  - Wichita Urology - Wichita Webb, Wichita, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic - Rochester Minnesota, Rochester, Minnesota
  - Minnesota Urology, Woodbury, Minnesota
  - The Urology Center, PC, Omaha, Nebraska
  - AMP UROLOGY, Syracuse - US Urology Partners, Syracuse, New York
  - SUNY Upstate Medical University Syracuse, Syracuse, New York
  - Montefiore Medical Center (Bronx2), The Bronx, New York
  - Central OH Urology Group - US Urology Partners, Gahanna, Ohio
  - Atlantic Urology Clinics - McLeod Health Blvd, Myrtle Beach, South Carolina
  - Urology Associates P C (Nashville), Nashville, Tennessee
  - University of Texas Southwestern Medical Center (Dallas), Dallas, Texas
  - University of Utah (Salt Lake City), Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Urology of Virginia (Virginia Beach), Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No